CLINICAL TRIAL: NCT03562000
Title: PReventing EXtubation FAILure by Cough Assistance and NIV in a Population Selected on Cough Peak Flow
Brief Title: PReventing EXtubation FAILure Related to Cough
Acronym: PREXFAIL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The primary evalution criteria had a so few occurrence that it has been a fundamental obstacle to randomize patient. The use of mecanical aide to cough is more widly employ, creating a second limitation.
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL18_0133
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Patients Intubated in ICU Before Extubation
Keywords: ICU; Cough; Randomised study; Cough assistance; Medical device; Physiotherapy
MeSH Terms: conditions — Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group on cough and ventilation assistance (Experimental): Mechanical cough assistance during physiotherapy post-extubation in ICU and systematic indication of NIV.
  Interventions: Device: Cough Assistance and Systematic Non-Invasive Ventilation
- Control group on cough and ventilation assistance (Other): Control group of extubated patients receiving the current gold standard strategy during physiotherapy after extubation in ICU and with selected indications of NIV.
  Interventions: Procedure: control group using the current gold standard of care after extubation, namely the manual drainage by a physiotherapist and the consensual use of Non-invasive ventilation

INTERVENTIONS:
Device: Cough Assistance and Systematic Non-Invasive Ventilation — A standardised bundle of intervention will be tested using the combination of two medical devices previously used in daily clinical practice but without guideline and objective selection criteria, namely:
  1. A mechanical cough assistance technic using the Cough Assist device (Model E70® by Philips Respironics, Carlsbad, CA, USA) before extubation then after extubation then 3 times a day (with possible additional treatment on demand) during 7 days maximum (with a possible cessation if the patient has strictly no bronchial overload during three consecutive physiotherapy sessions)
  2. A systematic Non-Invasive ventilation during 24h minimum to indirectly improve the clearance of bronchial overload and to reduce the overall risk of re-intubation related a relative hypoventilation associated to the weak cough.
  Arms: Intervention group on cough and ventilation assistance
Procedure: control group using the current gold standard of care after extubation, namely the manual drainage by a physiotherapist and the consensual use of Non-invasive ventilation — 1. After extubation, the physiotherapy will be managed according to standard care and cough assistance will be only manual. The use of a dedicated cough assistance device will be allowed if the bronchial overload clearance is repeatedly insufficient according to the physiotherapist in charge.
  2. Non-invasive ventilation will not be systematic and only used in case of pre-defined condition, such as: age > 65 years-old, BMI > 30, Chronic cardiac failure, COPD, hypercapnia at the end of the weaning trial, post-operative admissions after abdominal and thoracic surgery.
  Arms: Control group on cough and ventilation assistance

SUMMARY:
After the admission in ICU, most patients have to be intubated in order to control haematosis in case of acute respiratory failure, to reduce the metabolic crisis during severe haemodynamic shock, or to protect upper airways in case of impairment of consciousness. After the initial phase of etiological treatment, as soon as the patients no more required the intubation, weanibility has to be checked (thanks to a weaning trial with or without pressure support) before the separation attempt is decided on an evaluation of the overall extubability, based in particular on a subjective assessment of cough strength. The cases of re-intubation can be related to several factors such as: i) a ventilatory insufficiency indicating an imbalance between the muscular pomp function and the mechanical constraint of the chest; ii) an acute cardiogenic oedema; iii) an obstruction of the superior airways, possibly due to an imbalance between the bronchial overload and the cough efficacy.

Preventing extubation failure should avoid exposing such patients to an over-risk of morbidity and mortality due to the consequences of a prolonged invasive ventilation. This prevention can be implemented thanks to an early detection of the patients the most at risk and then a coherent intervention to manage of each risk factor involved. For example, the inspiratory insufficiency can be fixed by the use of Non-Invasive Ventilation (NIV), as proposed for patients developing a final hypercapnia at the end of the weanibility test.

Several studies have been conducted to improve the prediction of extubation failure. As this is notably influenced by the cough efficacy before extubation, it has been proposed to assess the peak flow expiratory during voluntary cough. The Cough Peak Flow could for example replaced some semi-quantitative measures of cough strength associated to a low reproducibility. The most validated threshold for a weak cough is < 60 L/min and it has recently been demonstrated that it remained valuable when directly assessed using the built-in ventilator flow-meter.

In the meantime, new devices of mechanical cough assistance have been developed and are frequently used for patients presenting a chronic neuro-muscular disease affecting their ability to spontaneously clear their airways from an inappropriate bronchial overload. However, the interest of such devices for a systematic use after extubation has not been validated with a sufficient level of evidence to be recommended, in particular because of the bias of the single randomised monocentric study.

The main objective of the study consists in demonstrating in an open multicentre randomised study (focused on the patients with an objective low cough strength) the superiority of a systematic strategy combining mechanical cough assistance and non-invasive ventilation on standard care (manual post-extubation physiotherapy and NIV for restrictive indications) to reduce the re-intubation rate at 48h.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years
2. Patients intubated for more than 24h before the extubation attempt
3. Patients able to follow simple commands (M6 response at the GCS) and to provide a signed agreement (or, in case of neurological impairment, to confirm to a third person their will to be included in the study by their appropriate code).
4. Successful weaning trial with a low pressure support (7 cmH2O) during 30-60 min or longer in case of neuromuscular disorders and with PEEP=0 cmH2O
5. Patients included for their first extubation attempt after a successful weaning trial based on classic weaning criteria (with the exception of: self-extubation, accidental extubation, extubation after less than 24 hours of ventilation).
6. No decision of care limitation on respiratory failure (reintubation considered).
7. Informed consent form signed by the patient (if cognitive capacities are preserved despite intubation) or by relatives (if cognitive and judgment capacities are impaired but with a capacity to respond to instructions sufficient to carry out spirometric measurements).
8. Randomisation if the cough is objectively assessed as weak (CPF < 60 L/min et VT < 0.55 L). In other case, the patient with a strong cough are only included in an observational study with an outcome assessment.

Exclusion Criteria:

1. Patient with tracheostomy
2. Weaning trial conducted without a pressure support technique during the last test
3. Failure of a weaning trial using a pressure support technique
4. Decision not to extubate after a successful weaning trial
5. Extubation of a patient already included after a previous extubation
6. Final extubation
7. Patients not affiliated to French health care system
8. Patients in poor medical condition (hemodynamic, respiratory instability)
9. Patients moribund or with previous decision of care limitation
10. Absence of informed consent document or patient under legal protection
11. Any clinical argument for a laryngeal oedema
12. No possibility of CPF assessment: ventilator non-adapted for assessment, no comprehension of the cough order despite a M6 response at the GCS (no coughing effort initiated).
13. Patient previously using a mechanical cough assistance
14. Deglutition disorders objectified or supposed (severe lesion of the brainstem), with a theoretical risk of tracheostomy
15. Contra-indication to mechanical cough assistance: pneumothorax or any lesion at risk of pneumothorax (such as costal fracture, emphysema, previous pneumothorax or other barotraumatism)
16. Contra-indication to Non-Invasive Ventilation: agitation, non-treated pneumothorax, thoracic wound, severe vomiting, active digestive haemorrhage with hematemesis, severe cranio-facial traumatism with pneumo-encephaly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Re-intubation rate, including every cause | 48 hours
  Re-intubation rate, including every causes evaluated at 48h (expressed as a percentage).
  The causes could including include cardiac arrest, acute haemodynamic failure, acute neurological failure (agitation or increased loss of wakefulness compared to the initial state), acute respiratory failure (clinical signs of ARF, namely increased breathing rate > 40/min, pH < 7.35, SpO2 < 92% during > 5 min using a Fi = 1, repeated desaturations, intolerance to Non Invasive Ventilation).
  Any death before 48h is considered as an extubation failure, whatever its cause.

SECONDARY OUTCOMES:
Evaluation of the efficacy on mortality. | 90 days or the duration of the hospitalisation.
  Assessing the mortality rate at 90 days post-randomisation/extubation and assessing complementarily the mortality rate at the ICU discharge and at the hospital discharge.
Evaluation of the efficiency on ICU care management | 90 days or the duration of the hospitalisation.
  Assessing the re-intubation rate at 7 days post-randomisation/extubation and assessing the overall extubation failure during the ICU hospitalisation (as a composite of the re-intubation rate and the tracheostomy rate). Describing the causes of re-intubation (related to bronchial overload, opposed to other causes such as acute pulmonary oedema, which will be analysed separately) and the post-extubation nosocomial pneumonia leading to a curative antibiotherapy in ICU. Assessing at 90 days post-randomisation/extubation the number of days without invasive respiratory support and without any respiratory support. Defining qualitatively the respiratory function at 90 days post-randomisation/extubation (dyspnoea, persistent bronchial overload, continuing physiotherapy). Describing the duration of: standard oxygenation, NIV after the first extubation, invasive ventilation after the first extubation, ICU stay and in-hospital stay.
Assessment of the clinical and biological efficacy of the cough assistance | 24 hours
  Comparing between the two groups: i) a semi-quantitatively evaluation of the bronchial overload before extubation and after the first physiotherapy treatment post extubation (with and without intervention, respectively) using a convenient "Bronchial Overload scale" build on a Likert basis defined between 1 (low bronchial overload with a better excepted extubation outcome) to 5 (high bronchial overload with a worse excepted extubation outcome) and assessed by an third party; ii) the difference of arterial blood gas (with and without mechanical intervention on cough, respectively).
Assessment of the clinical tolerance of the intervention | 7 days
  Assessing the number of treatment cessation due to tolerance issue and defined as Adverse Effects and Serious Adverse Effects. Describing the haemodynamic profiles of patient in both groups during the physiotherapy (with and without mechanical intervention on cough, respectively). Assessing the number of mechanical treatment failure requiring a change of the physiotherapy technique.

CONTACTS AND LOCATIONS:
Overall Officials: GOBERT Florent, MD, Study Director — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France